CLINICAL TRIAL: NCT03537287
Title: Intramuscular 17Alpha-hydroxyprogestrone, Progesterone Suppositories and Dydrogesterone Tablets in Preventing Preterm Labor
Brief Title: Different Types of Progesterone in the Prevention of Preterm Labor
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, mohammed mahmoud samy, Lecturer in Obstetrics and Gynecology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PDPTL
Record Dates: First submitted 2016-04-25; First posted 2018-05-25 (Actual); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Preterm Labor
MeSH Terms: conditions — Obstetric Labor, Premature | interventions — Dydrogesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 17 alpha hydroxyprogestrone caproate Group (Active Comparator): Patients will receive 250 mg of 17 alpha hydroxyprogestrone caproate intramuscularly once weekly starting from 16 weeks till delivery or 36 weeks.
  Interventions: Drug: 17 alpha hydroxyprogestrone caproate
- Vaginal progesterone Group (Active Comparator): Patients will receive vaginal progesterone 200 mg once per day starting from 16 weeks till delivery or 36 weeks.
  Interventions: Drug: Vaginal progesterone
- Oral dydrogesterone Group (Active Comparator): Patients will receive 2 tablets of oral dydrogesterone daily starting from 16 weeks till delivery or 36 weeks
  Interventions: Drug: Oral dydrogesterone

INTERVENTIONS:
Drug: 17 alpha hydroxyprogestrone caproate — 250 mg of 17 alpha hydroxyprogestrone caproate weekly
  Arms: 17 alpha hydroxyprogestrone caproate Group
Drug: Vaginal progesterone — 200 mg of vaginal progesterone daily
  Arms: Vaginal progesterone Group
Drug: Oral dydrogesterone — 2 tablets of dydrogesterone daily
  Arms: Oral dydrogesterone Group

SUMMARY:
Preterm birth is a common problem in obstetric care,with estimates ranging from 5% in several European countries to 18% in some African countries, Preterm labor defined as delivery before 37 completed weeks is the leading cause of perinatal and neonatal morbidity and mortality and strongly related to the developmental and neurological disabilities later in life..

There is still considerable uncertainty regarding the optimal progesterone type, route of administration, dosage and timing of start of therapy to prevent preterm labor in risky women

DETAILED DESCRIPTION:
This study aims to compare between the efficacy of intramuscular 17alpha-hydroxyprogestrone, progesterone vaginal suppositories and dydrogesterone oral tablets in prevention of preterm labor in high risk women.

All women will be counseled regarding mode of intervention and informed consent will be obtained. All cases will be subjected to complete history taking, routine antenatal examination and investigations, treatment of genital or urinary tract infections if diagnosed. Routine obstetric ultrasound examination and measurement of cervical length by transvaginal ultrasound will be carried out at 16-18weeks of pregnancy.

The study population will be randomly distributed according to the mode of intervention into 3 groups.

Randomization is performed using a Computer-generated randomization system. Blinding of the intervention is not feasible in this trial (owing to the different route of administration of the studied drugs).Table of randomization is obtained

Group 1:

Women who will take intramuscular 17 alpha hydroxyprogestrone caproate

Dose:

250 mg intramuscularly, once weekly starting from 16 weeks till delivery or 36 weeks.

Group 2 :

Women who will take progesterone 200mg vaginal suppositories.

Dose:

Once per day starting from 16 weeks till delivery or 36 weeks

Group 3 :

Women who will take oral dydrogesterone

Dose:

Take 2 tablets a day starting from 16 weeks till delivery or 36 weeks

Color Doppler blood flow velocity examination of fetal circulation will be performed by an independent investigator blinded to treatment before treatment &after two weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Living fetus with gestational age 16-18weeks (calculated according to date of last menstrual period confirmed with earlier ultrasound examination).
* Presence of risk factor for preterm labor:

  1. Previous spontaneous preterm labor in previous singleton Pregnancy, OR
  2. Previous spontaneous second trimestric miscarriage less than 3 times, OR
  3. Short cervix less than 25mm diagnosed during midtrimesteric transvaginal ultrasound examination at 16-18 weeks with or without history of previous preterm labor.

Exclusion Criteria:

* Multiple pregnancy.
* Medical or obstetric conditions requiring termination of pregnancy
* Contraindication to progesterone administration or its use earlier in this pregnancy

  * Current or past history of thrombophlebitis, thromboembolic disorders, or cerebral apoplexy.
  * Liver dysfunction or disease.
  * Known or suspected malignancy of breast or genital organs.
  * Undiagnosed vaginal bleeding.
  * Missed abortion.
  * Known sensitivity to progesterone injection.
  * Known sensitivity to sesame oil/seeds.
* Congenital fetal anomalies
* Cervical cerclage in the current pregnancy.
* Presence of uterine anomalies (Unicornuate uterus , Uterus didelphys, bicornuate uterus,Septated uterus) or uterine fibroid.
* Presence of history of chronic hypertetion, chronic liver or kidney diseases, and pregnancy induced hypertension.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Gestational age in weeks at delivery. | 6 months
  using either the last menstrual period in patients with regular cycles or early first trimester ultrasound to calculate the gestational age in weeks at delivery

SECONDARY OUTCOMES:
Hemodynamic changes in fetoplacental circulation | 6 months
  Measurement of U/S Doppler indices of umbilical artery and middle cerebral artery (namely PI, RI and S/D ratio) in fetal circulation
Unsatisfactory response | 6 months
  Number of patients who needed to increase the dose above the recommended initial dose.
Failure of prevention of preterm labor | 6 months
  Number of patients who suffered preterm labor and needed tocolysis
Birth weight | 6 months
  Birth weight in Kg
Neonatal APGAR score | 6 months
  Neonatal Apgar score at 1 and 5 min.
Need for NICU admission | 6 months
  Number of patients whose neonates were admitted to NICU
  Neonatal mortality.
Neonatal mortality | 6 months
  Number of neonatal deaths

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Samy, MD, Principal Investigator — M Samy
Locations (1):
- Ain SHams Maternity Hospital, Cairo, Abbaseya, Egypt

IPD SHARING:
Plan to Share IPD: No